CLINICAL TRIAL: NCT01245426
Title: A Phase II Randomised, Double-Blind, Placebo-Controlled, Parallel Group, Multicentre Study to Determine the Efficacy and Dose Response of Repeat Inhaled Doses of GW870086X on FEV1 in Adults With Persistent Asthma
Brief Title: A Study in Asthmatics to Determine the Efficacy and Dose Response of Repeat Doses of GW870086X on Forced Expiratory Volume in 1 Second (FEV1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114749
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Asthma; GW870086; Efficacy; FEV1
MeSH Terms: conditions — Asthma | interventions — GW870086X

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- GW870086 2mg (Experimental): GW870086 2mg once daily in the morning for 27 ± 2 days
  Interventions: Drug: GW870086 2mg
- GW870086 4mg (Experimental): GW870086 4mg once daily in the morning for 27 ± 2 days
  Interventions: Drug: GW870086 4mg
- Placebo (Placebo Comparator): Placebo once daily in the morning for 27 ± 2 days
  Interventions: Drug: GW870086 Placebo
- GW870086 1mg (Experimental): GW870086 1mg once daily in the morning for 27 ± 2 days
  Interventions: Drug: GW870086 1mg
- GW870086 3mg (Experimental): GW870086 3mg once daily in the morning for 27 ± 2 days
  Interventions: Drug: GW870086 3mg

INTERVENTIONS:
Drug: GW870086 2mg — oral inhalation
  Arms: GW870086 2mg
Drug: GW870086 4mg — oral inhalation
  Arms: GW870086 4mg
Drug: GW870086 Placebo — oral inhalation
  Arms: Placebo
Drug: GW870086 1mg — oral inhalation
  Arms: GW870086 1mg
Drug: GW870086 3mg — oral inhalation
  Arms: GW870086 3mg

SUMMARY:
This is a randomised, double-blind, placebo-controlled, parallel group study to determine the efficacy of twenty-seven day- repeat inhaled daily doses of GW870086X on forced expiratory volume in 1 second (FEV1). Initially there will be 3 treatment arms; placebo, 2mg GW870086X and 4mg GW870086X. After an interim analysis the trial may; continue to completion using the original doses, be terminated early, or have a fourth arm added of either 1mg GW870086X once daily or 3mg GW870086X once daily.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, parallel group study to determine the efficacy of twenty-seven day- repeat inhaled doses of GW870086X on FEV1. GW870086X is a novel inhaled corticosteroid with potent glucocorticoid activity currently in development by GlaxoSmithKline (GSK) as an inhaled treatment of persistent asthma. Initially, subjects will be randomised to receive placebo, 2mg or 4mg GW870086X once daily. An interim analysis will be performed on the primary endpoint to potentially adapt the study design after approximately 45 subjects have completed dosing. Based on the results of the interim analysis, the trial may continue to completion using the original doses or an adaptation to the doses could be made. Either the 1mg GW870086X once daily arm or 3mg GW870086X once daily arm may be added, or the trial could be terminated early. After screening there will be a 4 week run in period prior to start of treatment and after will be a follow up period 1-2 weeks after last dose. Approximately 120 subjects will complete the study. Key safety assessments include; clinical laboratory tests, vital signs and collection of adverse events (AE's).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years
* A female subject is eligible to participate if she is of: Non-childbearing potential. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.
* Male subjects must agree to use one of the protocol contraception methods.
* Body weight, men ≥ 50 kg, women ≥ 45 kg and BMI within the range 18.5 - 29.0 kg/m2 (inclusive).
* Documented history of bronchial asthma, first diagnosed at least 6 months prior to the screening visit and currently being treated only with intermittent short-acting beta-2 agonist therapy
* Severity of Disease: A best FEV1 of 60%-85% of the predicted normal value during the Visit 1 screening period.
* No history of smoking within 6 months of the start of the study and with a total pack year history of ≤10 pack years
* Capable of giving written informed consent
* Single QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* AST and ALT < 2xULN; alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* A positive test for Hepatitis B or Hepatitis C antibody.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* The subject has a positive pre-study drug/alcohol screen unless a positive can be explained by the patients' medication.
* Past or present disease, which as judged by the investigator, may affect the outcome of this study.
* Clinically significant abnormalities in safety laboratory analysis at screening, as determined by the investigator.
* Subject is hypertensive at screening.
* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnoea, respiratory arrest and/or hypoxic seizures.
* Administration of oral, injectable or dermal steroids within 8 weeks of screening.
* Exacerbation of asthma within 4 weeks prior to the first dose of study medication.
* Respiratory Infection that is not resolved within the 4 weeks before screening and led to a change in asthma management, or in the opinion of the Investigator is expected to affect the subjects asthma status or the subjects ability to participate in the study.
* Any asthma exacerbation requiring oral corticosteroids within 8 weeks of screening. A subject must not have had any hospitalisation for asthma within 6 months prior to screening
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. Paracetamol is an exception and will be permitted at daily doses of up to 4 g from screening to follow-up.
* Has taken Xanthines (including theophylline, but not including caffeine), anticholinergics, cromoglycates and/or long-acting beta-2 agonists within 1 week prior to screening and is unable to abstain from them throughout the study.
* Unable to abstain from other medications other than short acting inhaled beta-2 agonists and paracetamol (up to 4 g per day) 7 days before screening until the follow-up visit.
* Unable to abstain from medication or supplements that significantly inhibit the cytochrome P450 subfamily enzyme CYP3A4, from screening and throughout the study.
* Unable to use the DISKHALER® device correctly.
* History of sensitivity to any of the study medications.
* Where participation in the study would result in donation of blood or blood products in excess of 500 ml within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* The subject is not able to understand or comply with protocol requirements, instructions and protocol stated restrictions.
* Vulnerable subjects.
* Subject is mentally or legally incapacitated.
* Urinary cotinine levels indicative of smoking or history within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline associated with GW870086X versus placebo at Day 28 on FEV1 | Day 28

SECONDARY OUTCOMES:
Change from baseline in FEV1 on Day 7, Day 14 and Day 21 | Days; 7, 14, 21
Change from baseline in peak expiratory flow rate (PEFR) measured twice daily over 28 days | Days 1-28
Rescue medication usage | Days 1-28
Assessment of vital signs, safety laboratory parameters and incidences of adverse events throughout treatment period | 9-10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- GSK Investigational Site, Sofia, Bulgaria
- Germany (6):
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- South Africa (3):
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, George
  - GSK Investigational Site, Newton Park, Port Elizabeth

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114749 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114749 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114749 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114749 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114749 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114749 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114749 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register